CLINICAL TRIAL: NCT04655521
Title: The Dynamics of the Immune Response to Infection by SARS Coronavirus 2
Brief Title: Dynamics of the Immune Response to COVID-19 / Infection by SARS-CoV-2
Acronym: DIRECTOR
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Collaborators: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Principal Investigator, Cihan Papan, MD, Universität des Saarlandes
Other Study IDs: 109/20
Record Dates: First submitted 2020-12-02; First posted 2020-12-07 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; SARS-CoV-2; Viral Infection
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 patients
- Healthy controls
- Non-COVID-19 patients with respiratory tract infection

SUMMARY:
To evaluate host-immune biomarkers including TRAIL, IP-10, CRP and their computational integration for predicting COVID-19 and disease severity in patients with PCR-confirmed COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* confirmed infection with SARS-CoV-2 (except for the controls)

Exclusion Criteria:

* n/a

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects 3 months and older with suspicion of COVID-19 that present to the hospital due to suspected COVID-19. Controls with respiratory tract infection (Non-COVID-19) and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Differential expression of biomarkers between COVID-19 and controls | up to 90 days
  Differential expression of TRAIL, IP-10, CRP, and their computational integration in subjects with COVID-19, as compared to control subjects.
Differential expression of biomarkers between severe and non-severe COVID-19 | up to 90 days
  Differential expression of TRAIL, IP-10, CRP, and their computational integration in subjects with COVID-19, who require more extensive medical intervention (i.e., exhibit severe symptoms), i.e. severe infection vs. non-severe infection
Correlation of biomarkers with disease severity | up to 90 days
  Correlation between host-immune biomarkers including TRAIL, IP-10, CRP, and their computational integration for predicting disease severity in patients with COVID-19, where measures of severity include ICU admission, respiratory failure, mechanical ventilation, septic shock, non-respiratory organ failure, and mortality.

SECONDARY OUTCOMES:
Biomarkers depending on therapy | up to 90 days
  Differential expression of TRAIL, IP-10, CRP, and their computational integration in subjects with COVID-19 with or without specific therapy.
Biomarkers depending on bacterial co-infection | up to 90 days
  Differential expression of TRAIL, IP-10, CRP, and their computational integration in subjects with COVID-19 with or without bacterial co-infection.
Correlation of biomarkers with viral load | up to 90 days
  Correlation between host-immune biomarkers including TRAIL, IP-10, CRP, and their computational integration with infectiousness, i.e. e.g. viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Papan, MD, Principal Investigator — Universität des Saarlandes
Locations (1):
- Saarland University, Homburg, Germany

REFERENCES:
- [Background] Oved K, Cohen A, Boico O, Navon R, Friedman T, Etshtein L, Kriger O, Bamberger E, Fonar Y, Yacobov R, Wolchinsky R, Denkberg G, Dotan Y, Hochberg A, Reiter Y, Grupper M, Srugo I, Feigin P, Gorfine M, Chistyakov I, Dagan R, Klein A, Potasman I, Eden E. A novel host-proteome signature for distinguishing between acute bacterial and viral infections. PLoS One. 2015 Mar 18;10(3):e0120012. doi: 10.1371/journal.pone.0120012. eCollection 2015. PMID 25785720
- [Background] van Houten CB, de Groot JAH, Klein A, Srugo I, Chistyakov I, de Waal W, Meijssen CB, Avis W, Wolfs TFW, Shachor-Meyouhas Y, Stein M, Sanders EAM, Bont LJ. A host-protein based assay to differentiate between bacterial and viral infections in preschool children (OPPORTUNITY): a double-blind, multicentre, validation study. Lancet Infect Dis. 2017 Apr;17(4):431-440. doi: 10.1016/S1473-3099(16)30519-9. Epub 2016 Dec 22. PMID 28012942
- [Derived] Tegethoff SA, Danziger G, Kuhn D, Kimmer C, Adams T, Heintz L, Metz C, Reifenrath K, Angresius R, Mang S, Rixecker T, Becker A, Geisel J, Jentgen C, Seiler F, Reichert MC, Frohlich F, Meyer S, Rissland J, Ewen S, Wagenpfeil G, Last K, Smola S, Bals R, Lammert F, Becker SL, Krawczyk M, Lepper PM, Papan C. TNF-related apoptosis-inducing ligand, interferon gamma-induced protein 10, and C-reactive protein in predicting the progression of SARS-CoV-2 infection: a prospective cohort study. Int J Infect Dis. 2022 Sep;122:178-187. doi: 10.1016/j.ijid.2022.05.051. Epub 2022 May 25. PMID 35643306